CLINICAL TRIAL: NCT03282045
Title: A Multicenter, Single-blind, Randomized, Placebo-controlled Comparative Study on Efficacy and Safety of the Lysobact Complete Spray®, Tantum Verde® Spray and Pharyngal® Oromucosal Spray in the Treatment of Acute Sore Throat in Common Cold
Brief Title: Efficacy and Safety of the Lysobact Complete Spray®, Tantum Verde® and Pharyngal® Oromucosal Spray in the Treatment of Acute Sore Throat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bosnalijek D.D (Industry)
Collaborators: MonitorCRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BOS_CS_01
Record Dates: First submitted 2017-07-11; First posted 2017-09-13 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Sore Throat
Keywords: acute sore throat; lysobact
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lysobact Complete Sprey (Experimental): Lysobact Complete Sprey
  Route of administration: Oromucosal spray, sprayed directly toward the affected area with the applicator while the mouth is wide open
  Dose regimen: Sprayed 3 to 6 doses a day. For a single dose, spraying pump should be pressed 5 times and one press of the spray pump release 0.20 mL of the solution containing 4 mg lysozyme, 0.3 mg cetylpyridine and 0.1 mg lidocaine hydrochloride.
  Interventions: Drug: Lysobact Complete Sprey
- Tantum Verde® Spray (Active Comparator): Tantum Verde® Spray
  Route of administration: Oromucosal spray, sprayed directly toward the affected area with the applicator while the mouth is wide open.
  Dose regimen: Sprayed 4 to 8 doses, 2 to 6 times a day. One press means one dose.
  Interventions: Drug: Tantum Verde® Spray
- Pharyngal® Oromucosal Spray (Active Comparator): Pharyngal® Oromucosal Spray
  Route of administration: Oromucosal spray, sprayed directly toward the affected area with the applicator while the mouth is wide open.
  Dose regimen: Sprayed 2 to 4 doses, repeated 6 to 10 times per day. One press of the pump (one dose) releases 0.14 ml of the solution with 0.28 mg chlorhexidine digluconate and 0.07 mg of lidocaine hydrochloride.
  Interventions: Drug: Pharyngal® Oromucosal Spray
- Placebo (Placebo Comparator): Route of administration: Sprayed directly toward the affected area with the applicator while the mouth is wide open.
  Dose regimen: Sprayed 3 to 6 doses a day. For a single dose, spraying pump should be pressed 5 times.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lysobact Complete Sprey — Inhaling spray
  Arms: Lysobact Complete Sprey
Drug: Tantum Verde® Spray — Inhaling spray
  Arms: Tantum Verde® Spray
Drug: Pharyngal® Oromucosal Spray — Inhaling spray
  Arms: Pharyngal® Oromucosal Spray
Drug: Placebo — Inhaling spray
  Arms: Placebo

SUMMARY:
The primary objective of this multicenter, single-blind, randomized, placebo-controlled, prospective, comparative study with parallel design and 4-arms is to evaluate superiority of Lysobact Complete Spray® against placebo and non inferiority of Lysobact Complete Spray® against active comparators (Tantum Verde® and Pharyngal®) in terms of efficacy based on the pain VAS scores evaluated by the patient using Sore Throat Pain Intensity Scale (STPIS).

DETAILED DESCRIPTION:
This study will be conducted in approximately 3 centers in Bosnia Herzegovina and in 4 centers in Turkey.

Primary objective:

The primary objective of this study is to evaluate superiority of Lysobact Complete Spray® against placebo and non inferiority of Lysobact Complete Spray® against active comparators (Tantum Verde® and Pharyngal®) in terms of efficacy based on the pain VAS scores evaluated by the patient using Sore Throat Pain Intensity Scale (STPIS).

Secondary objective(s):

* Safety evaluation of Lysobact Complete Spray®, Tantum Verde® Spray, Pharyngal® Oromucosal Spray, based on the frequency and nature of adverse events occurring during treatment period.
* Extent of change in difficulty in swallowing, evaluated on the basis of Difficulty in Swallowing Scale (DSS), on Day 2, Day 4 and Day 6, as compared with baseline.
* Extent of change in swollen throat evaluation based on Swollen Throat Scale (STS) on Day 2, Day 4 and Day 6, as compared with baseline.
* Change in frequency of study treatment applications on Day 2, Day 4 and Day 6, as compared with baseline.

Test product: Lysobact Complete Spray® Active comparator product: Tantum Verde® Spray Active comparator product: Pharyngal® Oromucosal Spray Placebo product: Placebo

Primary endpoint:

• Primary endpoint is the change from baseline to Day 6 in mean VAS score for STPIS.

Secondary endpoint(s):

Secondary endpoints are as follows:

* change from baseline to Day 6 in mean VAS score for DSS
* change from baseline to Day 6 in mean VAS score for SwoTS
* change from baseline to each visit (Day 2, Day 4, Day 6) for STPIS , DSS and SwoTS
* percent improvement from baseline to each visit (Day 2, Day 4, Day 6) for STPIS , DSS and SwoTS
* Incidence of adverse events and relationship to the study treatments
* Incidence of serious adverse events and relationship to the study treatments

Statistical methods:

All patients who have received at least one dose of any study medication will be included in the safety evaluation (safety population). Patients who have completed all visits according to the protocol will be included in the efficacy population. The superiority and inferiority of Lysobact Complete Spray® will be tested in hierarchical order by the comparison of the mean change of VAS scores [Sore Throat Pain Intensity Scale (STPIS)] from baseline to Day 2, 4 and 6.

Planned treatment duration is 5 days. Safety will be followed-up until Day 6. End of study is defined as the end of the follow up period for the last patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute tonsillo-pharyngitis symptoms in common cold and by using a scale-based symptom Tonsillo-Pharyngitis Assessment (TPA) as an objective finding of pharyngeal infection, with a score of ≥5
* Patients who will be treated only on a symptomatic treatment basis, and with a prescribed a oropharyngeal spray
* Patients, 18 years of age and above, who provided an informed consent
* Patients with a sore-throat of recent onset, symptoms initiated ≤48 hours
* Patients with sore throat pain rated ≥66 mm on the Sore Throat Pain Intensity Scale (STPIS)
* Patients with difficulty in swallowing rated ≥50 mm on Difficulty Swallowing Scale (DSS)
* Patients with a sensation of swollen throat rated ≥33 mm on the Swollen Throat Scale (SwoTS)

Exclusion Criteria:

* Patients who had any previous (within 4 hours prior to screening examination) throat lozenge treatment/use
* Patients who had used any flu-preparation which contains any analgesic ingredient such as paracetamol, ibuprofen or acetylsalicylic acid (ASA) along with a decongestant
* Patients who had analgesic use (any) 4 hours prior to the screening examination
* Patients who are prescribed an antibiotic use before the screening visit and are entitled to use antibiotics during the course of this non-interventional study
* Patients with a known hypersensitivity to active/inactive ingredients of medications which is prescribed for the symptomatic treatment of sore throat
* Patients with known hypersensitiveness to egg white and other allergens
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2016-10; Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
to evaluate superiority of Lysobact Complete Spray® against placebo and non-inferiority of Lysobact Complete Spray® against active comparators | Day 6
  The primary objective of this study is to evaluate superiority of Lysobact Complete Spray® against placebo and non-inferiority of Lysobact Complete Spray® against active comparators (Tantum Verde® and Pharyngal®) in terms of efficacy based on the pain VAS scores evaluated by the patient using Sore Throat Pain Intensity Scale (STPIS).

CONTACTS AND LOCATIONS:
Overall Officials: OZGUN ENVER, MD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- University Clinical Center of the Republic of Srpska, ENT Clinic, Banja Luka, Bosnia and Herzegovina, Banja Luka, Bosnia and Herzegovina